CLINICAL TRIAL: NCT04786275
Title: Evaluation of the Nociception Guided by NoL Index and Pharmacokinetics of Fentanyl in Pediatric Patients Under General Anesthesia for Non-cardiac Elective Surgery
Brief Title: Evaluation of the Nociception Guided by NoL Index and PK of Fentanyl in Pediatric Patients Under General Anesthesia
Acronym: NoLPedFenta
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Francisco Cruzat, Principal Investigator, Pontificia Universidad Catolica de Chile
Other Study IDs: 190416008
Record Dates: First submitted 2021-01-27; First posted 2021-03-08 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Pain; Anesthesia; Pediatric ALL
Keywords: NoL; Nociception level; Fentanyl; Pediatric anesthesia; Pharmacokinetics
MeSH Terms: conditions — Pain; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tetanic stimulation: Single arm study
  Interventions: Drug: Fentanyl; Other: Tetanic stimulation

INTERVENTIONS:
Drug: Fentanyl — Standard dose of 2 ug/kg after tetanic stimulation.
Other: Tetanic stimulation — Standard tetanic stimulation will be used as the stimulus to evaluate response of the intraoperative pain index (NoL) at a standard fentanyl dose.

SUMMARY:
Fentanyl is one of the most common used opioids for analgesia during general anesthesia, however there are few studies that describe the relationship between its pharmacokinetics and pharmacodynamics, especially in the pediatric population. The monitoring of the analgesia component during general anesthesia has been traditionally by changes in patient's vital signs, with new devices that measure nociceptive indexes like the Nociception level (NoL) index currently being validated for adults. There is still lacking evidence with nociceptive indexes in the pediatric population.

Insufficient dose of opioids may cause sympathetic response, respiratory complications, development of persistent post-surgical pain and even prolonged hospitalization. In the other hand, and overdose of opioids may cause over sedation, postoperatory nausea and vomiting, respiratory depression, hyperalgesia and tolerance.

Given the lack of evidence on the Pharmacokinetic and pharmacodynamic (PK/PD) of fentanyl in this group of patients, has led to raise the development of this observational prospective study; which is to describe a PK/PD model of fentanyl in pediatric population, through evaluation of the NoL index, in patients submitted to elective general non-cardiac surgery.

DETAILED DESCRIPTION:
Patients will be invited to participate before surgery, the inclusion criteria will be revised and the informed consent will be signed by one of the parents or legal tutor.

In the operating room will be recorded demographic data and relevant background such as: Age, Weight, Size, BMI.

Afterwards, in the operating room, the patient will be monitored regularly: EKG, pulse oximetry, non invasive blood pressure.

Induction of anesthesia with sevoflurane 6% in 100% oxygen, once loss of consciousness, 2 peripheral IV lines will be installed, one for medication and the other in the contralateral arm for blood samples. After that, a laryngeal mask device (LMA) appropriate for the weight for the management of the airway. In addition, the EEG will be monitored through a frontal electroencephalographic monitoring (BIS) system and a NoL index sensor, both of which will be recorded throughout the surgery.

Once all monitors are installed, a caudal block with 0,5-1 ml of bupivacaine 0,25% will be performed, in the left decubitus lateral position. Ventilator and vaporizer adjustments for an EtCO2 of 35-40 mmHg and a BIS index of 50-60 with Sevoflurane. After 12 minutes, because of the latency of caudal block; surgeons may start. If an effective caudal block is proven, the study will continue; if there is movement of the child, laryngospasm or an increase of more than 10% in the base values of heart rate or blood pressure, the patient will be excluded from the study.

Standardized nociceptive stimulus will be administered through a tetanic stimulus (70 Hz, 80 mA) for 5 seconds in the forearm. An initial tetanic stimulus will be performed, 2 minutes afterwards a unique dose of fentanyl of 2 micrograms per kg will be administered. New tetanic stimulus will be applied at 5, 15, 30 and 45 minutes after the fentanyl dose and blood samples for fentanyl plasmatic levels will be taken at the same time in the operating room and at 75 or 120 minutes in the post anesthesia care unit (PACU). NoL index values will be recorded after each tetanic stimulus.

After surgery, sevoflurane will be discontinued, LMA removed and the patients transferred to the PACU. Pain scores will be evaluated in the PACU using Visual analogue scale. Analgesic management with NSAIDs and Acetaminophen.

PK/PD profile of fentanyl will be evaluated with NONMEM (non-linear mixed effects modelling) software for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-10 years old
* ASA I - II
* Lower abdominal or urological surgery, requiring general anesthesia and caudal block

Exclusion Criteria:

* Obese patients
* ASA III - IV - V
* Allergy to fentanyl
* Emergency surgery
* Patients with sleep apnea
* Surgeries anticipated to have an increased volume exchange or transfusion

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ASA I or II children from 3 up to 10 years requiring elective non-cardiac surgery, under general anesthesia and caudal block.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
NoL index. | Since induction of anesthesia until emergence of anesthesia (one hour in average)
  Variations in the NoL index (0-100). NoL has a range from 0-100, with 0 indicates no pain and 100 indicates worst pain. Data will also be analyzed using nonlinear mixed effect modeling (NONMEM)
Change of the plasmatic levels of fentanyl | 5, 15, 30, 45, 75 until 120 minutes after one dose of fentanyl.
  Describe the change of the levels of fentanyl plasmatic levels (ng/mL) measured by high pressure liquid chromatography (HPLC).
Peak Plasma Concentration (Cmax) | 5, 15, 30, 45, 75 until 120 minutes after one dose of fentanyl.
  Calculate maximum plasma concentration (Cmax) fentanyl plasma levels measured with high pressure fluid (HPLC) after a single bolus of fentanyl in enrolled pediatric patients.

SECONDARY OUTCOMES:
Hemodynamics | At time of surgery, up to 120 minutes.
  Arterial pressure (mmHg)
Heart rate (bpm) | At time of surgery, up to 120 minutes
  Heart rate (bpm)
Pulse oximetry | At time of surgery, up to 120 minutes.
  % oximetry saturation
Bispectral index | At time of surgery, up to 120 minutes
  Depth of anesthesia will be recorded with BIS monitor
Pain in Visual analogue scale (0-10) | Every 15 minutes in the PACU, up to 120 minutes
  Postoperative pain will be evaluated with Visual analogue scale (0-10), being a score of 10 worst outcome, in the PACU for 120 minutes immediately after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Pedemonte, MSc, MD, Study Director — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Analysis plan

REFERENCES:
- [Background] Ziesenitz VC, Vaughns JD, Koch G, Mikus G, van den Anker JN. Pharmacokinetics of Fentanyl and Its Derivatives in Children: A Comprehensive Review. Clin Pharmacokinet. 2018 Feb;57(2):125-149. doi: 10.1007/s40262-017-0569-6. PMID 28688027
- [Background] Lotsch J. Pharmacokinetic-pharmacodynamic modeling of opioids. J Pain Symptom Manage. 2005 May;29(5 Suppl):S90-103. doi: 10.1016/j.jpainsymman.2005.01.012. PMID 15907650
- [Background] Renaud-Roy E, Stockle PA, Maximos S, Brulotte V, Sideris L, Dube P, Drolet P, Tanoubi I, Issa R, Verdonck O, Fortier LP, Richebe P. Correlation between incremental remifentanil doses and the Nociception Level (NOL) index response after intraoperative noxious stimuli. Can J Anaesth. 2019 Sep;66(9):1049-1061. doi: 10.1007/s12630-019-01372-1. Epub 2019 Apr 17. PMID 30997633